CLINICAL TRIAL: NCT01368640
Title: Generation of Prediction Equations to Analyze Body Composition of Adults Based on Bioelectrical Impedance Analysis (BIA)
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-01
Record Dates: First submitted 2011-04-15; First posted 2011-06-08 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Bioelectrical Impedance Measurement of Healthy Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy adults: The study will cover 130 healthy adults. 65 men and 65 women in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.

SUMMARY:
Aim of the study is to develop prediction equations for calculating FFM, TBW, ECW and SMM based on the gold standard reference methods ADP, DXA, MRI, D2O and NaBr on the one hand and measurement data of the BIA devices on the other hand. The equations are necessary to use the device as a Body Composition Analyzer with an acceptable accuracy level for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

The study will cover 130 healthy adults. 65 men and 65 women in an age range of 18 to 65 years with a BMI of 18.5 to 35 kg/m2 are planned to be recruited.

Exclusion Criteria:

* acute and chronic diseases
* regular intake of medications (except for contraceptives)
* amputation of limbs
* electrical implant as cardiac pacemaker
* insulin pumps
* artificial joints
* metallic implants (except tooth implants)
* claustrophobia
* pregnancy or breastfeeding period
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the inv. site
* current alcohol abuse
* frequent hypersensitivity reactions/allergies determ. anamnestically
* body weight of more than 150 kg
* extensive tattoos at arms or legs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data of 130 healthy adults are planned to be collected.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bioelectrical Impedance of 5 and 50 kHz for one body side | 15 minutes
Bioelectrical Impedance of 50 kHz for all 4 extremities | 15 minutes

SECONDARY OUTCOMES:
Bioelectrical Impedance of 1, 1.5, 2, 3, 7.5, 10, 15, 20, 30, 75, 100, 150, 200, 300, 500, 750 and 1,000 kHz | 15 minutes
  The measurement is planned to be done for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side. In total resistance and reactance at 19 frequencies for 7 body segments are planned to be measured.
Generation of prediction equations for Sceletal Muscle Mass based on MRI | 1 hour
Bioelectrical Impedance in sitting, lying and standing | 15 minutes
Precision Study | 15 min
  The precision study pursues three targets:
  1. Repeatability (variability across successive measurements within a short time period taken by the same operator and the same device; device is repositioned between successive measurements).
  2. Between-operator precision (variability across measurements taken by the same device, but different operators).
  3. Between-device precision (variability across measurements taken by the same operator, but different devices).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred J. Mueller, Prof. Dr. med., Principal Investigator — Christian-Albrechts-University of Kiel
Locations (1):
- Institute of Human Nutrition and Food Science, Kiel, Germany

REFERENCES:
- [Derived] Enderle J, Reljic D, Jensen B, Peine S, Zopf Y, Bosy-Westphal A. Normal values for body composition in adults are better represented by continuous reference ranges dependent on age and BMI. Clin Nutr. 2023 May;42(5):644-652. doi: 10.1016/j.clnu.2023.03.006. Epub 2023 Mar 9. PMID 36933351
- [Derived] Jensen B, Braun W, Both M, Gallagher D, Clark P, Gonzalez DL, Kluckmann K, Bosy-Westphal A. Configuration of bioelectrical impedance measurements affects results for phase angle. Med Eng Phys. 2020 Oct;84:10-15. doi: 10.1016/j.medengphy.2020.07.021. Epub 2020 Jul 30. PMID 32977906